CLINICAL TRIAL: NCT03523390
Title: A Phase I/Ib Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of Avelumab in Chinese Subjects With Locally Advanced Unresectable or Metastatic Solid Tumors With Expansion to Selected Indication(s)
Brief Title: Phase I/Ib Multiple Ascending Dose Study in China
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: MS100070_0035
Record Dates: First submitted 2018-05-01; First posted 2018-05-14 (Actual); Results first posted 2024-02-23 (Actual); Last update posted 2024-02-23 (Actual); Status verified 2023-07

CONDITIONS: Metastatic Solid Tumors
Keywords: Metastatic Solid Tumors; Avelumab; MSB0010718C
MeSH Terms: interventions — avelumab

STUDY DESIGN:
Intervention Model Description: Subsequent cohorts of subjects treated at different dose levels in this study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Avelumab 3 mg/kg Q2W (Experimental)
  Interventions: Drug: Avelumab 3 mg/kg Q2W
- Avelumab 10 mg/kg Q2W (Experimental)
  Interventions: Drug: Avelumab 10 mg/kg Q2W
- Avelumab 20 mg/kg Q2W (Experimental)
  Interventions: Drug: Avelumab 20 mg/kg Q2W
- Avelumab 10 mg/kg QW (Experimental)
  Interventions: Drug: Avelumab 10 mg/kg QW

INTERVENTIONS:
Drug: Avelumab 3 mg/kg Q2W — Participants received intravenous infusion of Avelumab over 1 hour duration at a dose of 3 milligrams per kilogram (mg/kg) once every 2 weeks (Q2W) until disease progression, significant clinical deterioration, unacceptable toxicity, or any criterion for withdrawal from the study or from Avelumab occurs.
  Other Names: MSB0010718C
  Arms: Avelumab 3 mg/kg Q2W
Drug: Avelumab 10 mg/kg Q2W — Participants received intravenous infusion of Avelumab over 1 hour duration at a dose of 10 mg/kg Q2W until disease progression, significant clinical deterioration, unacceptable toxicity, or any criterion for withdrawal from the study or from Avelumab occurs.
  Arms: Avelumab 10 mg/kg Q2W
Drug: Avelumab 20 mg/kg Q2W — Participants received intravenous infusion of Avelumab over 1 hour duration at a dose of 20 mg/kg Q2W until disease progression, significant clinical deterioration, unacceptable toxicity, or any criterion for withdrawal from the study or from Avelumab occurs.
  Arms: Avelumab 20 mg/kg Q2W
Drug: Avelumab 10 mg/kg QW — Participants received intravenous infusion of Avelumab over 1 hour duration at a dose of 10 mg/kg every week (QW) for the first 12 weeks followed by once every 2 weeks, started at Week 13 until disease progression, significant clinical deterioration, unacceptable toxicity, or any criterion for withdrawal from the study or from Avelumab occurs.
  Arms: Avelumab 10 mg/kg QW

SUMMARY:
The purpose of this study was to evaluate the maximum tolerated dose (MTD) and pharmacokinetics (PK) of Avelumab monotherapy in Chinese subjects.

ELIGIBILITY:
Inclusion Criteria:

* Signed written informed consent prior to any study-related procedures are undertaken that are not part of standard patient management
* Histologically or cytologically proven locally advanced unresectable or metastatic solid tumors, for which no standard therapy exists or standard therapy has failed
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1 at study entry
* Availability of a recently obtained formalin-fixed, paraffin-embedded block containing tumor tissue (biopsy from a non-irradiated area within 6 months) or 12 or more unstained tumor slides suitable for biomarker detection
* Other protocol defined inclusion criteria could apply

Exclusion Criteria:

* Prior therapy with any antibody/drug targeting T-cell coregulatory proteins (immune checkpoints) such as programmed death 1 (PD-1), PD-L1, cytotoxic T-lymphocyte antigen-4 (CTLA-4), 4-1BB, Lymphocyte-activation gene 3 (LAG-3), T-cell immunoglobulin and mucin-domain containing-3 (TIM-3) or anti-Cluster of Differentiation (CD)-127
* Persisting toxicity related to prior therapy (Grade greater than equals to [>=] 2 National Cancer Institute- Common Terminology Criteria for Adverse Events [NCI-CTCAE] v4.03, except Grade less than [<] 3 neuropathy and alopecia of any grade)
* Concurrent anticancer treatment (for example, cytoreductive therapy, radiotherapy [with the exception of limited palliative bone-directed radiotherapy], immune therapy, or cytokine therapy except for erthyropoietin).
* Concurrent immunosuppressive agents (except for corticosteroids at physiologic replacement dose, equivalent to less than equals to [<=] 10 milligram [mg] prednisone daily)
* Severe hypersensitivity reactions to monoclonal antibodies (Grade >= 3 NCI-CTCAE v4.03)
* Active brain metastases (except those treated locally, and have not been progressing for at least 2 weeks after the completion of therapy, with no steroid maintenance therapy required, and no ongoing neurological symptoms related to brain localization of the disease)
* Any history of anaphylaxis, or uncontrolled asthma (that is, 3 or more features of partially controlled asthma)
* Other protocol defined exclusion criteria could apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2018-04-24 (Actual); Primary Completion 2019-07-29 (Actual); Study Completion 2021-02-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director — Merck KGaA, Darmstadt, Germany
Locations (3):
- China (3):
  - Research site, Guangzhou, Guangzhou
  - Research site, Changchun, Jilin
  - Research site, Hangzhou, Zhejiang

REFERENCES:
- [Result] Wu YL, Cheng Y, Chen H, Tu H, Xu C, Wang Z, Liu Y, Xin Y, Lou H, Wang W, Chin K, Li D, Zhao D, Gao Y, Xu W, Pan H. Phase I/Ib dose-escalation study of avelumab in Chinese patients with advanced solid tumors. Future Oncol. 2022 Jun;18(17):2053-2062. doi: 10.2217/fon-2021-1342. Epub 2022 Mar 31. PMID 35354274
- See also: Trial Awareness and Transparency website — https://clinicaltrials.emdgroup.com/en/trial-details/?id=MS100070_0035
- See also: Medical Information Location Map - Med Info Contacts — https://www.merckgroup.com/en/company/contact-us/medinfo-contact-map.html

RESULTS

PARTICIPANT FLOW:
Groups:
- Avelumab 10 mg/kg Q2W: Participants received intravenous infusion of Avelumab over 1 hour duration at a dose of 10 mg/kg once Q2W until disease progression, significant clinical deterioration, unacceptable toxicity, or any criterion for withdrawal from the study or from Avelumab occurs.
- Avelumab 20 mg/kg Q2W: Participants received intravenous infusion of Avelumab over 1 hour duration at a dose of 20 mg/kg once Q2W until disease progression, significant clinical deterioration, unacceptable toxicity, or any criterion for withdrawal from the study or from Avelumab occurs.
- Avelumab 10 mg/kg QW: Participants received intravenous infusion of Avelumab over 1 hour duration at a dose of 10 mg/kg once every week (QW) for the first 12 weeks followed by once every 2 weeks, started at Week 13 until disease progression, significant clinical deterioration, unacceptable toxicity, or any criterion for withdrawal from the study or from Avelumab occurs.
Period: Overall Study
Arm/Group | Avelumab 3 mg/kg Q2W | Avelumab 10 mg/kg Q2W | Avelumab 20 mg/kg Q2W | Avelumab 10 mg/kg QW
Started | 3 | 7 | 6 | 8
Completed | 3 | 7 | 6 | 8
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety analysis set (SAF) included all participants who have received at least 1 dose of Avelumab.
Groups:
- Total: Total of all reporting groups
Arm/Group | Avelumab 3 mg/kg Q2W | Avelumab 10 mg/kg Q2W | Avelumab 20 mg/kg Q2W | Avelumab 10 mg/kg QW | Total
Number analyzed (Participants) | 3 | 7 | 6 | 8 | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 54 (17.7) | 52 (14.3) | 50 (16.6) | 61 (13.1) | 55 (14.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 2 | 4 | 4 | 10
  Male | 3 | 5 | 2 | 4 | 14
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 3 | 7 | 6 | 8 | 24
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With of Dose-limiting Toxicities (DLTs) According to National Cancer Institute Common Toxicity Criteria for Adverse Events (NCI-CTCAE) Version 4.03
Description: DLT is defined as greater than or equal to [>=] Grade (Gr)3 Adverse drug reaction (ADR) according to NCI-CTCAE v4.03, occurring during DLT observation period of dose escalation cohorts. ADR: any AE suspected to be related to avelumab by Investigator and/Sponsor. Following events were not considered as DLT: Gr3 infusion-related reaction resolving within 6 hours and controlled with medical management. Transient (less than or equal to [<=] 6 hours) Gr3 flu-like symptoms/fever, controlled with medical management. Transient (<=24 hours) Gr3 fatigue, local reactions, headache, nausea, emesis, resolves to <= Gr1. Gr3 skin toxicity/Gr3 Liver function test increase that resolves to <= Grade 1 in < 7 days after medical management. Gr3 diarrhea, out-of-range laboratory values without any clinical correlate that resolves to <= Grade 1 within 7 days with adequate medical management; Tumor flare phenomenon defined as local pain, irritation, rash localized at sites of known or suspected tumor.
Time Frame: Day 1 to Day 21
Population: DLT analysis set included all participants with data used for implementing the dose escalation schedule (excluding 6 participants in 10 mg/kg once weekly cohort) and received all Avelumab administrations in the DLT observation period or should have stopped treatment because of DLTs in the DLT observation period.
Measure: Count of Participants; unit: Participants
Arm/Group | Avelumab 3 mg/kg Q2W | Avelumab 10 mg/kg Q2W | Avelumab 20 mg/kg Q2W
Number analyzed (Participants) | 3 | 7 | 3
Participants | 0 | 0 | 0

2. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs) and Treatment Related TEAEs According to National Cancer Institute- Common Terminology Criteria for Adverse Events Version 4.03 (NCI-CTCAE v4.03)
Description: An Adverse event (AE) was defined as any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease associated with the use of study drug, whether or not considered related to the study drug or worsening of pre-existing medical condition, whether or not related to study drug. A serious adverse event (SAE) was an AE that resulted in any of the following outcomes: death; life threatening; persistent/significant disability/incapacity; initial or prolonged inpatient hospitalization; congenital anomaly/birth defect or was otherwise considered medically important. TEAEs were defined as events that emerge during treatment having been absent pre-treatment, or worsen relative to the pre-treatment state and with onset dates occurring within the first dosing day of study treatment until 30 days after the last dose of study treatment. TEAEs include both Serious TEAEs and non-serious TEAEs. Treatment-related TEAEs: reasonably related to the study intervention.
Time Frame: Time from first study treatment up to 139 weeks
Population: SAF included all participants who have received at least 1 dose of Avelumab.
Measure: Count of Participants; unit: Participants
Arm/Group | Avelumab 3 mg/kg Q2W | Avelumab 10 mg/kg Q2W | Avelumab 20 mg/kg Q2W | Avelumab 10 mg/kg QW
Number analyzed (Participants) | 3 | 7 | 6 | 8
Participants
  Participants with TEAEs | 3 | 7 | 6 | 8
  Participants with Treatment Related TEAEs | 3 | 6 | 6 | 6

3. Secondary Outcome: Number of Participants With at Least 1 Positive Anti-Avelumab Antibodies (ADA)
Description: Serum samples were analyzed by a validated electrochemiluminescence immunoassay to detect the presence of antidrug antibodies (ADA). Number of participants with ADA positive results for Avelumab were reported.
Time Frame: Time from first study treatment up to 139 weeks
Population: Immunogenicity Analysis Set included all participants who have any dose of avelumab and who have at least one valid ADA result.
Measure: Count of Participants; unit: Participants
Arm/Group | Avelumab 3 mg/kg Q2W | Avelumab 10 mg/kg Q2W | Avelumab 20 mg/kg Q2W | Avelumab 10 mg/kg QW
Number analyzed (Participants) | 3 | 7 | 6 | 8
Participants | 2 | 0 | 0 | 0

4. Primary Outcome: Area Under the Serum Concentration Time Curve From Time Zero to the Time of the Last Quantifiable Concentration (AUC0-t) of Avelumab
Description: Area under the serum concentration-time curve from time zero to the last sampling time at which the concentration is at or above lower limit of quantification (LLOQ). AUC0-t was calculated according to the mixed log linear trapezoidal rule.
Time Frame: Day 1: within 2 hours prior to and at the end of the 1-hour infusion, and at 0.5, 1, 2, 4, 6, and 12 hours after the end of the infusion
Population: Pharmacokinetics (PK) analysis set included all participants who have completed at least 1 infusion of avelumab, and who have provided valid PK samples. As pre-specified in statistical analysis plan (SAP), data for AUC0-t was planned to be reported for Avelumab 3 mg/kg Q2W, Avelumab 10 mg/kg Q2W and Avelumab 20 mg/kg Q2W arms only.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram*hour per milliliter (mcg*h/mL)
Arm/Group | Avelumab 3 mg/kg Q2W | Avelumab 10 mg/kg Q2W | Avelumab 20 mg/kg Q2W
Number analyzed (Participants) | 3 | 7 | 6
microgram*hour per milliliter (mcg*h/mL) | 7000 (3.0) | 20400 (31.3) | 35600 (20.6)

5. Primary Outcome: Area Under the Serum Concentration-Time Curve During a Dosing Interval (AUCtau) of Avelumab
Description: AUCtau was defined as area under the serum concentration-time curve from time zero to the end of the dosing interval (tau). AUCtau was calculated using the mixed log linear trapezoidal rule.
Time Frame: as for outcome 4
Population: PK analysis set included all participants who have completed at least 1 infusion of avelumab, and who have provided valid PK samples. As pre-specified in SAP, data for AUCtau was planned to be reported for Avelumab 3 mg/kg Q2W, Avelumab 10 mg/kg Q2W and Avelumab 20 mg/kg Q2W arms only.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mcg*h/mL
Arm/Group | Avelumab 3 mg/kg Q2W | Avelumab 10 mg/kg Q2W | Avelumab 20 mg/kg Q2W
Number analyzed (Participants) | 3 | 7 | 6
mcg*h/mL | 7000 (2.9) | 20800 (27.8) | 35800 (22.3)

6. Primary Outcome: Area Under the Serum Concentration-Time Curve From Time Zero Extrapolated to Infinity (AUC0-inf) of Avelumab
Description: AUC0-inf was calculated by combining AUC0-t and AUCextra. AUCextra represents an extrapolated value obtained by Clast pred/Lambda z, where Clast pred was the calculated serum concentration at the last sampling time point at which the measured serum concentration is at or above the Lower Limit of quantification (LLOQ) and Lambda z was the apparent terminal rate constant determined by log-linear regression analysis of the measured serum concentrations of the terminal log-linear phase.
Time Frame: as for outcome 4
Population: PK analysis set included all participants who have completed at least 1 infusion of avelumab, and who have provided valid PK samples. As pre-specified in SAP, data for AUC0-inf was planned to be reported for Avelumab 3 mg/kg Q2W, Avelumab 10 mg/kg Q2W and Avelumab 20 mg/kg Q2W arms only.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mcg*h/mL
Arm/Group | Avelumab 3 mg/kg Q2W | Avelumab 10 mg/kg Q2W | Avelumab 20 mg/kg Q2W
Number analyzed (Participants) | 3 | 7 | 6
mcg*h/mL | 7710 (6.2) | 22600 (29.7) | 38300 (23.4)

7. Primary Outcome: Terminal Elimination Rate Constant (Lambda z) of Avelumab
Description: Lambda z was determined from the terminal slope of the log-transformed serum concentration curve using linear regression method.
Time Frame: as for outcome 4
Population: PK analysis set included all participants who have completed at least 1 infusion of avelumab, and who have provided valid PK samples. As pre-specified in SAP, data for Lambda z was planned to be reported for Avelumab 3 mg/kg Q2W, Avelumab 10 mg/kg Q2W and Avelumab 20 mg/kg Q2W arms only.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: 1/hour
Arm/Group | Avelumab 3 mg/kg Q2W | Avelumab 10 mg/kg Q2W | Avelumab 20 mg/kg Q2W
Number analyzed (Participants) | 3 | 7 | 6
1/hour | 0.00719 (18.6) | 0.00767 (21.1) | 0.00811 (9.1)

8. Primary Outcome: Maximum Observed Serum Concentration (Cmax) of Avelumab
Description: Cmax was obtained directly from the serum concentration versus time curve.
Time Frame: as for outcome 4
Population: PK analysis set included all participants who have completed at least 1 infusion of avelumab, and who have provided valid PK samples. As pre-specified in SAP, data for Cmax was planned to be reported for Avelumab 3 mg/kg Q2W, Avelumab 10 mg/kg Q2W and Avelumab 20 mg/kg Q2W arms only.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram per milliliter (mcg/mL)
Arm/Group | Avelumab 3 mg/kg Q2W | Avelumab 10 mg/kg Q2W | Avelumab 20 mg/kg Q2W
Number analyzed (Participants) | 3 | 7 | 6
microgram per milliliter (mcg/mL) | 77.6 (13.9) | 294 (44.7) | 450 (36.5)

9. Primary Outcome: Last Quantifiable Serum Concentration (Clast) of Avelumab
Description: Clast is the last measurable serum concentration of Avelumab.
Time Frame: as for outcome 4
Population: PK analysis set included all participants who have completed at least 1 infusion of avelumab, and who have provided valid PK samples. As pre-specified in SAP, data for Clast was planned to be reported for Avelumab 3 mg/kg Q2W, Avelumab 10 mg/kg Q2W and Avelumab 20 mg/kg Q2W arms only.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mcg/mL
Arm/Group | Avelumab 3 mg/kg Q2W | Avelumab 10 mg/kg Q2W | Avelumab 20 mg/kg Q2W
Number analyzed (Participants) | 3 | 7 | 6
mcg/mL | 4.94 (33.7) | 16.3 (51.2) | 21.4 (50.3)

10. Primary Outcome: Serum Trough Concentration Levels (Ctrough) of Avelumab
Description: Ctrough is defined as the concentration observed immediately before next dosing.
Time Frame: Day 1: within 2 hours prior to 1 hour infusion
Population: PK analysis set included all participants who have completed at least 1 infusion of avelumab, and who have provided valid PK samples. Here, "Overall Number of Participants Analyzed" signifies those participants who were evaluable for this outcome measure. As pre-specified in SAP, data for Ctrough was planned to be reported for Avelumab 3 mg/kg Q2W, Avelumab 10 mg/kg Q2W and Avelumab 20 mg/kg Q2W arms only.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mcg/mL
Arm/Group | Avelumab 3 mg/kg Q2W | Avelumab 10 mg/kg Q2W | Avelumab 20 mg/kg Q2W
Number analyzed (Participants) | 3 | 6 | 6
mcg/mL | 4.94 (33.7) | 14.8 (47.2) | 21.4 (50.3)

11. Primary Outcome: Time to Reach Maximum Observed Serum Concentration (Tmax) of Avelumab
Description: The time to reach the maximum observed serum concentration (tmax) was obtained directly from the concentration versus time curve.
Time Frame: as for outcome 4
Population: PK analysis set included all participants who have completed at least 1 infusion of avelumab, and who have provided valid PK samples. As pre-specified in SAP, data for tmax was planned to be reported for Avelumab 3 mg/kg Q2W, Avelumab 10 mg/kg Q2W and Avelumab 20 mg/kg Q2W arms only.
Measure: Median (Full Range); unit: hours
Arm/Group | Avelumab 3 mg/kg Q2W | Avelumab 10 mg/kg Q2W | Avelumab 20 mg/kg Q2W
Number analyzed (Participants) | 3 | 7 | 6
hours | 1.55 [1.53 to 1.62] | 1.52 [1.00 to 6.90] | 1.97 [1.05 to 5.00]

12. Primary Outcome: Apparent Terminal Half Life (t1/2) of Avelumab
Description: Apparent terminal half-life was defined as the time required for the serum concentration of drug to decrease 50 percent in the final stage of its elimination. t1/2 was calculated as log2/ lambda z. Lambda z was determined from the terminal slope of the log-transformed serum concentration curve using linear regression method.
Time Frame: as for outcome 4
Population: PK analysis set included all participants who have completed at least 1 infusion of avelumab, and who have provided valid PK samples. As pre-specified in SAP, data for t1/2 was planned to be reported for Avelumab 3 mg/kg Q2W, Avelumab 10 mg/kg Q2W and Avelumab 20 mg/kg Q2W arms only.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | Avelumab 3 mg/kg Q2W | Avelumab 10 mg/kg Q2W | Avelumab 20 mg/kg Q2W
Number analyzed (Participants) | 3 | 7 | 6
hours | 96.5 (18.6) | 90.3 (21.1) | 85.5 (9.1)

13. Primary Outcome: Dose Normalized Area Under the Serum Concentration-Time Curve From Time Zero to the Last Sampling Time (AUC0-t/Dose) of Avelumab
Description: AUC0-t/Dose was defined as area under the serum concentration versus time curve from time of dosing to the time of the last measurable concentration divided by dose. AUC0-t/Dose was measured in (microgram*hour per milliliter)/(milligram per kilogram) (mcg*h/mL)/(mg/kg).
Time Frame: as for outcome 4
Population: PK analysis set included all participants who have completed at least 1 infusion of avelumab, and who have provided valid PK samples. As pre-specified in SAP, data for AUC0-t/dose was planned to be reported for Avelumab 3 mg/kg Q2W, Avelumab 10 mg/kg Q2W and Avelumab 20 mg/kg Q2W arms only.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: (mcg*h/mL)/(mg/kg)
Arm/Group | Avelumab 3 mg/kg Q2W | Avelumab 10 mg/kg Q2W | Avelumab 20 mg/kg Q2W
Number analyzed (Participants) | 3 | 7 | 6
(mcg*h/mL)/(mg/kg) | 2330 (3.0) | 2040 (31.3) | 1780 (20.6)

14. Primary Outcome: Dose Normalized Area Under the Concentration-Time Curve Over the Dosing Interval (AUCtau/Dose) of Avelumab
Description: AUCtau/Dose was calculated by as dose normalized area under the serum concentration-time curve from time zero to the end of the dosing interval (tau). AUCtau was calculated using the mixed log linear trapezoidal rule.
Time Frame: as for outcome 4
Population: PK analysis set included all participants who have completed at least 1 infusion of avelumab, and who have provided valid PK samples. As pre-specified in SAP, data for AUCtau/dose was planned to be reported for Avelumab 3 mg/kg Q2W, Avelumab 10 mg/kg Q2W and Avelumab 20 mg/kg Q2W arms only.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: (mcg*h/mL)/(mg/kg)
Arm/Group | Avelumab 3 mg/kg Q2W | Avelumab 10 mg/kg Q2W | Avelumab 20 mg/kg Q2W
Number analyzed (Participants) | 3 | 7 | 6
(mcg*h/mL)/(mg/kg) | 2330 (2.9) | 2080 (27.8) | 1790 (22.3)

15. Primary Outcome: Dose Normalized Maximum Observed Serum Concentration (Cmax/Dose) of Avelumab
Description: Cmax/Dose was defined as maximum observed serum concentration divided by dose.
Time Frame: as for outcome 4
Population: PK analysis set included all participants who have completed at least 1 infusion of avelumab, and who have provided valid PK samples. As pre-specified in SAP, data for Cmax/dose was planned to be reported for Avelumab 3 mg/kg Q2W, Avelumab 10 mg/kg Q2W and Avelumab 20 mg/kg Q2W arms only.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: (mcg/mL)/(mg/kg)
Arm/Group | Avelumab 3 mg/kg Q2W | Avelumab 10 mg/kg Q2W | Avelumab 20 mg/kg Q2W
Number analyzed (Participants) | 3 | 7 | 6
(mcg/mL)/(mg/kg) | 25.9 (13.9) | 29.4 (44.7) | 22.5 (36.5)

ADVERSE EVENTS:
Time Frame: Time from first study treatment up to 139 weeks
Arm/Group | Avelumab 3 mg/kg Q2W | Avelumab 10 mg/kg Q2W | Avelumab 20 mg/kg Q2W | Avelumab 10 mg/kg QW
All-Cause Mortality (participants affected / at risk) | 1/3 | 4/7 | 6/6 | 7/8
Serious Adverse Events (participants affected / at risk) | 1/3 | 3/7 | 2/6 | 2/8
Other Adverse Events (participants affected / at risk) | 3/3 | 7/7 | 6/6 | 8/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Avelumab 3 mg/kg Q2W (N=3) | Avelumab 10 mg/kg Q2W (N=7) | Avelumab 20 mg/kg Q2W (N=6) | Avelumab 10 mg/kg QW (N=8)
Anemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Hepatic failure (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 1 | 0
Head injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 1
Hyperuricemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Apnea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Bronchostenosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Avelumab 3 mg/kg Q2W (N=3) | Avelumab 10 mg/kg Q2W (N=7) | Avelumab 20 mg/kg Q2W (N=6) | Avelumab 10 mg/kg QW (N=8)
Anaemia (Blood and lymphatic system disorders) | 2 | 4 | 6 | 6
Neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Atrioventricular block first degree (Cardiac disorders) | 1 | 0 | 0 | 0
Atrioventricular block second degree (Cardiac disorders) | 1 | 0 | 0 | 0
Bundle branch block right (Cardiac disorders) | 0 | 0 | 0 | 1
Sinus arrhythmia (Cardiac disorders) | 0 | 0 | 1 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 1 | 1 | 1
Supraventricular tachycardia (Cardiac disorders) | 0 | 1 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 2 | 0 | 0
Ventricular extrasystoles (Cardiac disorders) | 1 | 0 | 0 | 0
Autoimmune thyroiditis (Endocrine disorders) | 0 | 0 | 0 | 1
Hypothyroidism (Endocrine disorders) | 0 | 0 | 1 | 1
Vision blurred (Eye disorders) | 0 | 2 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 1 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Ascites (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 2 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 2
Epigastric discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 1 | 4
Vomiting (Gastrointestinal disorders) | 0 | 1 | 1 | 1
Asthenia (General disorders) | 0 | 1 | 0 | 0
Chest discomfort (General disorders) | 0 | 1 | 0 | 2
Chest pain (General disorders) | 0 | 3 | 1 | 1
Chills (General disorders) | 1 | 1 | 0 | 0
Fatigue (General disorders) | 1 | 1 | 1 | 1
Feeling cold (General disorders) | 0 | 0 | 1 | 0
Influenza like illness (General disorders) | 0 | 1 | 0 | 0
Malaise (General disorders) | 0 | 1 | 2 | 0
Non-cardiac chest pain (General disorders) | 1 | 0 | 0 | 1
Oedema peripheral (General disorders) | 0 | 1 | 0 | 0
Pain (General disorders) | 0 | 0 | 0 | 1
Pyrexia (General disorders) | 1 | 2 | 3 | 4
Swelling face (General disorders) | 0 | 0 | 0 | 1
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 1
Gingivitis (Infections and infestations) | 0 | 0 | 0 | 1
Herpes zoster (Infections and infestations) | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 1 | 1
Skin infection (Infections and infestations) | 0 | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Activated partial thromboplastin time prolonged (Investigations) | 0 | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 1 | 2 | 1
Amylase increased (Investigations) | 0 | 1 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 2 | 1
Bilirubin conjugated increased (Investigations) | 0 | 2 | 0 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 3 | 0 | 1
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 2
Blood chloride increased (Investigations) | 0 | 0 | 0 | 1
Blood creatinine increased (Investigations) | 0 | 2 | 1 | 2
Blood lactate dehydrogenase increased (Investigations) | 0 | 0 | 0 | 1
Blood phosphorus increased (Investigations) | 0 | 0 | 0 | 1
Blood pressure increased (Investigations) | 0 | 0 | 1 | 0
Blood thyroid stimulating hormone decreased (Investigations) | 0 | 0 | 1 | 1
Blood urea increased (Investigations) | 0 | 1 | 0 | 0
Electrocardiogram QT prolonged (Investigations) | 0 | 2 | 1 | 1
Gamma-glutamyltransferase increased (Investigations) | 0 | 2 | 2 | 1
Heart rate increased (Investigations) | 0 | 0 | 0 | 1
International normalised ratio increased (Investigations) | 0 | 0 | 0 | 1
Low density lipoprotein increased (Investigations) | 0 | 0 | 1 | 0
Lymphocyte count decreased (Investigations) | 0 | 1 | 2 | 0
Neutrophil count decreased (Investigations) | 0 | 0 | 0 | 1
Platelet count decreased (Investigations) | 0 | 0 | 1 | 1
Prothrombin time prolonged (Investigations) | 0 | 0 | 0 | 1
Red blood cells urine positive (Investigations) | 0 | 2 | 0 | 0
Reticulocyte count increased (Investigations) | 0 | 2 | 0 | 0
Urinary sediment present (Investigations) | 0 | 1 | 0 | 0
Urine output decreased (Investigations) | 0 | 0 | 0 | 1
Weight decreased (Investigations) | 2 | 5 | 2 | 4
Weight increased (Investigations) | 0 | 1 | 0 | 0
White blood cells urine positive (Investigations) | 0 | 3 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 3 | 2 | 3
Glycopenia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1
Hypernatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 3 | 0 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 2 | 2 | 2
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Hypochloraemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 3 | 0 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hypoproteinaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Lactic acidosis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Metabolic acidosis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 1 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Neck mass (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Aphasia (Nervous system disorders) | 0 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 2 | 3
Dysgeusia (Nervous system disorders) | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 0 | 1 | 0 | 2
Syncope (Nervous system disorders) | 0 | 1 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 1 | 1 | 2
Dysuria (Renal and urinary disorders) | 0 | 0 | 0 | 1
Haematuria (Renal and urinary disorders) | 0 | 2 | 0 | 1
Proteinuria (Renal and urinary disorders) | 1 | 3 | 2 | 3
Oedema genital (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Pelvic fluid collection (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Bronchostenosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 1 | 1
Dry throat (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 3
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 2
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 2 | 2
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2 | 0
Sputum discoloured (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Dermatitis bullous (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Leukoderma (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Vitiligo (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Yellow skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Bedridden (Social circumstances) | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-05-17): https://cdn.clinicaltrials.gov/large-docs/90/NCT03523390/Prot_000.pdf
  • Statistical Analysis Plan (2019-08-13): https://cdn.clinicaltrials.gov/large-docs/90/NCT03523390/SAP_001.pdf